CLINICAL TRIAL: NCT01384435
Title: A Randomized, Double Blind, Placebo-controlled Phase II Study of KPS-0373 in Patients With SCD
Brief Title: A Phase II Double Blind Comparative Study of KPS-0373 in Patients With Spinocerebellar Degeneration (SCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KPS1203
Record Dates: First submitted 2011-06-23; First posted 2011-06-29 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-03

CONDITIONS: SCD
Keywords: Spinocerebellar degeneration (SCD); Thyrotropin-Releasing Hormone (TRH)
MeSH Terms: conditions — Spinocerebellar Degenerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- KPS-0373, lowest dose (Experimental)
  Interventions: Drug: KPS-0373
- KPS-0373, 2nd lowest dose (Experimental)
  Interventions: Drug: KPS-0373
- KPS-0373, 2nd highest dose (Experimental)
  Interventions: Drug: KPS-0373
- KPS-0373, highest dose (Experimental)
  Interventions: Drug: KPS-0373
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KPS-0373
  Arms: KPS-0373, lowest dose
Drug: KPS-0373
  Arms: KPS-0373, 2nd lowest dose
Drug: KPS-0373
  Arms: KPS-0373, 2nd highest dose
Drug: KPS-0373
  Arms: KPS-0373, highest dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KPS-0373 compared to placebo in patients with Spinocerebellar Degeneration (SCD).

ELIGIBILITY:
Inclusion Criteria:

* Japanese SCD patients with mild to moderate ataxia

Exclusion Criteria:

* Patients with secondary ataxia
* Patients with clinically significant hepatic, renal, or cardiovascular dysfunction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Scale for the assessment and rating of ataxia (SARA) | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in patient improvement impression of activities of daily living | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katsumi Hontani, Study Director — Clinical Research Dept.
Locations (1):
- Japan, Tokyo and Other Japanese City, Japan